CLINICAL TRIAL: NCT05371041
Title: Defining Targets for Tic Detection and Suppression in Tourette Syndrome Deep Brain Stimulation
Brief Title: Tourette Deep Brain Stimulation (DBS) Target Detection & Suppression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB202102161; UH3NS119844 (NIH); OCR41251 (Other: UFOnCore)
Record Dates: First submitted 2022-05-06; First posted 2022-05-12 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Medtronic Percept Neurostimulator (Experimental): This is a deep brain stimulator that can also record brain signals and deliver stimulation through a control algorithm based on brain activity.
  Interventions: Device: Medtronic Percept Neurostimulator

INTERVENTIONS:
Device: Medtronic Percept Neurostimulator — This is a deep brain stimulator that can also record brain signals and deliver stimulation through a control algorithm based on brain activity.

SUMMARY:
The investigators will implant and monitor 8 research subjects with a subcortical closed-loop system for detection and suppression of tics in subjects with medically refractory debilitating Tourette Syndrome. The project will use the FDA-approved "Medtronic Percept PC" device, which is an implantable neurostimulator capable of recording neural signals. The study will target the CM nucleus of the thalamus and the aGPi in each brain hemisphere from each subject and we will connect the two leads placed in each brain hemisphere to two Percept devices.

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a continuous lifelong condition that is highly prevalent, socially disabling, and in some severe cases, physically injurious. Deep Brain Stimulation (DBS) has emerged as a promising treatment option for addressing uncontrollable tics in medically refractory, severe cases of TS frequently involving self-injurious behavior. We have undertaken a major informatics initiative by establishing the International TS DBS Registry and Database, a multi-country consortium that has captured long term outcomes of 277 TS DBS patients representing 50-75% of all TS DBS cases worldwide. From these outcomes, two deep brain targets have emerged as potentially effective: the centromedian nucleus region (CM) of the thalamus, and the anterior globus pallidus internus (aGPi). However, our current understanding of tic generation is limited by many factors including a lack of animal models for TS, apparently normal brain structure on structural imaging, and the impracticality of studying involuntary motor tics with functional imaging. Next generation closed-loop DBS systems can record brain activity in patients with TS and identify the neurophysiological correlates of tics. Moreover, these devices can deliver stimulation in response to a patient's symptomatic state. Our overall goal is to develop neurophysiology driven and connectivity-guided closed-loop DBS systems for the improved treatment of TS. To this end, we will implant 8 medically resistant TS patients with bilateral leads in the CM and aGPi. In Aim 1, we will identify structural network projections from CM and aGPi to guide pre-operative surgical planning and post-operative selection of stimulation parameters. In Aim 2, we will identify neurophysiologic correlates of tic genesis in the CM and aGPi. We will also study thalamo-pallidal network interactions leading to and during tics. In Aim 3, we will test the feasibility, safety, and efficacy of closed-loop TS DBS. We expect that closed-loop stimulation will provide more effective and personalized treatment options with longer battery life and fewer adverse effects than traditional chronic stimulation.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of TS must be made by both a fellowship-trained movement disorders neurologist and a psychiatrist and must meet Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for a diagnosis of TS.
* Yale Global Tic Severity Scale (YGTSS; 100) must be >35/50 and the motor tic sub score >15. The TS must be causing incapacitation with severe distress, self-injurious behavior, and/or quality of life disruption. OCD, Depression, and ADHD are not exclusionary provided tics are the major difficulty requiring surgical intervention.
* There are no gender criteria for this study.
* The subject's TS symptoms must be medication refractory. To meet the medication refractory criteria, subjects must have been treated by a psychiatrist or neurologist experienced in TS with therapeutic doses (doses adapted from Scahill's recommendations of at least three dopamine blocking drugs) [either 1-4 mg/day of haloperidol, 2-8 mg/day of pimozide, risperidone (1-3 mg/day), or aripiprazole (2.5-5 mg/day)]. There must be at a minimum7 single trial with an alpha-2 adrenergic agonist (0.1-0.3 mg/day).
* Clinically relevant depression if present must be pharmacologically treated and deemed stable (by the study psychiatrist).
* Must have been stabilized for one month on TS medication without a dose change prior to surgical intervention. If medication trials resulted in discontinuation of TS medications, the subject must be stabilized for three months off TS medicines.
* Must be willing to keep TS related medications stable and unchanged throughout the trial.
* Must have been offered habit reversal therapy/cognitive behavioral intervention therapy (HRT) if a subject did not have it prior to enrollment. Subjects are not required to participate in HRT but it will be highly encouraged, and must be completed prior to the start of the protocol. Those who improve significantly with HRT will be excluded from receiving surgery.
* If the tic is focal or addressable by botulinum toxin treatment, the study neurologist will offer to administer a trial of botulinum toxin prior to consideration of surgical therapy. If the subject chooses not to have the treatment, they cannot participate in the study. If the subject responds satisfactorily to botulinum toxin, and their quality of life significantly improves, they will be excluded from the study.
* Must be 18 years of age or older.8

Exclusion Criteria:

* • Any previous neurosurgical intervention such as DBS or ablative brain lesions. Participants with previous DBS system that have been explanted will still be excluded from the study.

  * Any metal in the body that would preclude the patient from receiving an MRI scan.
  * Untreated or unstable anxiety, depression, bipolar disorder or other Axis I psychiatric disorder.
  * Presence of psychotic features.
  * Significant psychosocial factors that may impart an increased risk.
  * The presence of only simple motor tics, a movement disorder other than TS, or medication related movement disorders from TS medications.
  * The presence of drug-induced tics (potentially associated with the use of stimulant medications, anticonvulsant drugs, etc.).
  * Severe medical co-morbidity including cardiovascular disorder, lung disorder, kidney disease, chronic neurological disease, hematological disease, or frailty that impact tolerability of the surgery as judged by the screening physicians.
  * Abnormal brain magnetic resonance imaging (MRI) scan including hydrocephalus, stroke, structural lesions, demyelinating lesions, or infectious lesions that would potentially confound the outcome or safety of the surgery as judged by the study neurosurgeon. Also excluded if severe atrophy is present on the brain scan.
  * Dementia or cognitive dysfunction that will place the subject at risk for worsening cognition, and/or may impact the ability to cooperate with tasks involved in the study.
  * Any attempt or intent of suicide in the last six months.
  * Significant substance abuse or dependence (e.g., stimulants, alcohol, opiates, benzodiazepines) within the past six months.
  * A positive urine drug screen for illicit substances (a urine drug screen is required), not to include marijuana/cannabinoid use.
  * Patients who do not have access to a site that can program the device if they cannot come to The University of Florida for clinical re-programming follow-up appointments after completion of the study.
  * Multiple failed medication treatments of inadequate dose or duration.
  * History of noncompliance with previous medical and psychosocial treatment efforts.
  * Severe head banging tics (any tics which have the potential to result in damage to the DBS as judged by the neurosurgeon).
  * Women of child-bearing potential who are pregnant or who wish to become pregnant during the study (a urine pregnancy screen required).
  * History of multiple surgical procedures with poor outcomes.
  * Unexplained gaps in medical history.
  * Pending lawsuits or other legal action.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale_(YGTSS) - Total Tic Score | 9 months
  The YGTSS is a clinician-rated scale used to assess tic severity over the prior week. It includes a checklist of motor and vocal tics followed by an assessment of the number, frequency, intensity, complexity, and inference of motor tics and phonic tics - scored separately. Each of these dimensions is scored on a 0 to 5 scale. The YGTSS provides three tic severity scores: Total Motor (0 to 25); Total Phonic (0 to 25) and the combined Total Tic Severity Score (0 to 50), as well as a separate Impairment dimension scored from 0 to 50. The Total Tic Score (YGTSS-TTS) was used in these analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Okun, MD, Principal Investigator — University of Florida; Christopher Butson, PhD, Principal Investigator — University of Florida; Aysegul Gunduz, PhD, Principal Investigator — University of Florida
Locations (1):
- Norman Fixel Institute for Neurological Diseases - University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No